CLINICAL TRIAL: NCT01659801
Title: Clinical Evaluation of the Toric BuunyLens TR Intra-ocular Lens
Brief Title: Evaluation of the BunnyLens TR Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BunnyLens TR 70 EMS
Record Dates: First submitted 2012-08-01; First posted 2012-08-08 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cataract
Keywords: cataract; cataract surgery; intaocular lens; toric lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BunnyLens TR — BunnyLens TR IOL is an Aspheric Toric intraocular lens providing a precise, superior alternative to surgical treatment of pre-existing corneal astigmatism.
  Other Names: toric inta-ocular lens

SUMMARY:
With age, a human crystalline lens opacifies (cataract) disabling the eye in generating a clear, well contrasted image. The only therapeutic solution to this problem is surgical replacement of the crystalline lens with an intraocular lens (cataract surgery).

In addition to the cataract, the person might suffer from pre-existing cormeal astigmatism. In cases of severe corneal astigmatism, the standard IOL might not provide the optimal result, and additional surgical procedures as Incisional Keratotomy or Limbal Relaxing Incisions might be required.

BunnyLens TR IOL is an Aspheric Toric intraocular lens providing a precise, superior alternative to surgical treatment of pre-existing corneal astigmatism.

The BunnyLens TR IOL is designed for micro-incision cataract surgery (MICS), through 1.8mm incisions.

The aims of this study are to:

* Demonstrate a reduction in refractive cylinder compared to pre-operative corneal astigmatism
* Exceed monocular best corrected distance visual acuity results provided in ISO guidelines.

DETAILED DESCRIPTION:
The reduction in refractive cylinder compared to pre-operative corneal astigmatism will be assessed using pre- and postoperative subjective refraction evaluation. Units of the measurement: diopters.

Monocular best corrected distance visual acuity will be assessed using ETDRS charts. Units of the measurement: logMAR.

There are no complications related to the BunnyLens TR implantation beyond those that might be expected in standard cataract surgery. The complications will be reported using Ocular condition forms included in the CRFs.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 years of age, of either gender and any race;
* Have preoperative corneal astigmatism of >= 2 Dpt as determined by IOL Master keratometry;
* Have regular, bowtie shaped corneal astigmatism. Corneal topography printout should be approved and signed by cornea specialist.
* Anterior chamber depth is between 2.5 to 3.8 mm
* Axial length is between 22 to 26 mm
* are willing and able to understand and sign an informed consent;
* have age related cataracts that require extraction followed by implantation of a posterior chamber intraocular lens (IOL) and used as an on-label procedure;
* are able to obtain pupil dilation >=4.0 mm.

Exclusion Criteria:

* Following disease(s)/condition(s): choroidal hemorrhage, chronic severe uveitis, concomitant severe eye disease, microphthalmos, proliferative diabetic retinopathy, corneal dystrophy, optic nerve atrophy, uncontrolled glaucoma or glaucoma treated by 3 or more medications, uncontrolled systemic disease or any ocular condition, that by opinion of investigator would compromise the refractive outcome or potential of the eye to achieve good vision.
* High intraocular pressure (above 25mmHg)
* Previous intraocular or corneal surgery;
* Corneal abnormality that would prevent stable and reliable visual acuity and refractive measures;
* Current rigid contact lens usage (within 3 months prior to the preoperative biometry reading)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
monocular best corrected distance visual acuity results 3 months after BunnyLens TR implantation | 3 months
• Demonstrate a reduction in refractive cylinder compared to pre-operative corneal astigmatism | 3 months

SECONDARY OUTCOMES:
Complications related to BunnyLens TR implantation duting cataract surgery | 3 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Lang, MD, Principal Investigator — Ha'Emek Medical Center, Afula Israel